CLINICAL TRIAL: NCT00014560
Title: Phase I Trial Of Intravenous Bispecific Antibody (4G7XH22) In Patients With Refractory Or Relapsed Non-Hodgkin's Lymphoma Or Chronic Lymphocytic Leukemia (CLL)
Brief Title: Antibody Therapy in Treating Patients With Refractory or Relapsed Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Medarex (supplier of BsAb) stopped study due to toxicities experienced at other sites on unrelated trials halting manufacturing of BsAb
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068556; P30CA023108 (NIH); DMS-9806; NCI-G01-1936
Record Dates: First submitted 2001-04-10; First posted 2003-07-30 (Estimated); Results first posted 2013-08-05 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Leukemia; Lymphoma
Keywords: refractory chronic lymphocytic leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell | interventions — Antibodies, Bispecific; sargramostim

ARMS (1):
- Single arm (Experimental): Antibody
  Interventions: Biological: bispecific antibody 4G7xH22; Biological: sargramostim

INTERVENTIONS:
Biological: bispecific antibody 4G7xH22
Biological: sargramostim

SUMMARY:
RATIONALE: Antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of antibody therapy in treating patients who have refractory or relapsed non-Hodgkin's lymphoma or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of bispecific antibody 4G7xH22 in patients with relapsed or refractory non-Hodgkin's lymphoma or chronic lymphocytic leukemia.
* Assess the clinical toxicity of this antibody in these patients.

OUTLINE: This is a dose escalation study of bispecific antibody (BsAb) 4G7xH22.

Patients receive sargramostim (GM-CSF) subcutaneously on day 1 and BsAb 4G7xH22 IV over 2 hours on day 2. Treatment repeats weekly for a total of 3 courses in the absence of unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BsAb 4G7xH22 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 6 patients experience dose-limiting toxicity.

Patients are followed weekly for 4 weeks, monthly for 3 months, and then periodically for 1 year.

PROJECTED ACCRUAL: Approximately 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of CD19+ non-Hodgkin's lymphoma or chronic lymphocytic leukemia

  * Primary refractory or multiply relapsed (after at least 2 prior chemotherapy regimens) disease
  * Ineligible for bone marrow or peripheral blood stem cell transplantation

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* Alkaline phosphatase less than 2 times normal
* SGPT less than 2 times normal

Renal:

* Creatinine clearance greater than 50 mL/min

Other:

* No human-anti-murine-antibody response to prior murine monoclonal antibodies
* No immunological or inflammatory disease (e.g., lupus erythematosus)
* No active serious infection
* No other serious medical condition that would limit survival to less than 2 years
* No other active malignancy except non-melanoma skin cancer or carcinoma in situ of the cervix
* No psychiatric or addictive disorder that would preclude study
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior immunotherapy allowed

Chemotherapy:

* See Disease Characteristics
* No concurrent chemotherapy

Endocrine therapy:

* Concurrent steroids for adrenal failure or adverse reactions to study drug allowed
* Concurrent hormonal therapy for non-disease related conditions (e.g., insulin for diabetes) allowed

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2000-09-28 (Actual); Primary Completion 2003-02-14 (Actual); Study Completion 2003-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Ely, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: This is a Phase 1a/1b trial. three patients will be treated at dose level 1.If no Grade 3 or 4 toxicities, the next dose level will be given to a new cohort of three. If 1 of 3 patients suffer Grade 3 or 4 toxicity, an additional 3 patients will be treated at same dose level.if 1/6 have a Grade 3 or 4 toxicity, proceed to next dose level with a cohort of 3 patients. If > 1/6 experience garde 3 or 4 toxicity, the DLT has been reached and the MTD is the dose level prior. Six patients will be treated at the MTD.
Period: Overall Study
Arm/Group | Single Arm
Started | 3
Completed | 0
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Clinical Toxicity
Description: This study was prematurely ended by the sponsor Medarex (supplier of BsAb) due to toxicities experienced at other sites on unrelated trials leading to the decision that Medarex would not be manufacturing the investigational product (BsAb).
Time Frame: day 1-29
Population: This study was prematurely ended by the sponsor Medarex (supplier of BsAb) due to toxicities experienced at other sites on unrelated trials leading to the decision that Medarex would not be manufacturing the investigational product (BsAb).
Arm/Group | Single Arm
Number analyzed (Participants) | 0

2. Primary Outcome: Determine the Maximum Tolerated Dose (MTD) and Dose Limiting Toxicity (DLT) of BsAb 4G7 x 22
Description: as for outcome 1
Time Frame: Day 1-29
Reporting Status: Not Posted

3. Secondary Outcome: Serum Markers of Macrophage Activation
Description: as for outcome 1
Time Frame: Day 1 Hours 0,2,4,6,24, day 15 Hours 0,2,4,6,24
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
This study was prematurely ended by the sponsor Medarex (supplier of BsAb) due to toxicities experienced at other sites on unrelated trials leading to the decision that Medarex would not be manufacturing the investigational product (BsAb).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes